CLINICAL TRIAL: NCT00005606
Title: Adoptive Immunotherapy of Epstein Barr Virus Induced Lymhoproliferative Disease. A Comparison of Allogeneic and Autologous Lymphocyte Responses ex Vivo and Use of Highly Selected Reactive Cells as an Alternative to Chemotherapy in Vivo.
Brief Title: Peripheral Blood Lymphocyte Therapy to Prevent Lymphoproliferative Disorders Caused by Epstein-Barr Virus in Patients Who Have Undergone Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: NU 98H1; NU-98H1; NCI-G00-1739
Record Dates: First submitted 2000-05-02; First posted 2003-01-27 (Estimated); Last update posted 2012-06-06 (Estimated); Status verified 2012-05

CONDITIONS: Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm
Keywords: stage I adult Hodgkin lymphoma; stage II adult Hodgkin lymphoma; stage III adult Hodgkin lymphoma; stage IV adult Hodgkin lymphoma; recurrent childhood acute lymphoblastic leukemia; recurrent adult Hodgkin lymphoma; stage I cutaneous T-cell non-Hodgkin lymphoma; stage II cutaneous T-cell non-Hodgkin lymphoma; stage III cutaneous T-cell non-Hodgkin lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; isolated plasmacytoma of bone; extramedullary plasmacytoma; stage 0 chronic lymphocytic leukemia; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; stage I chronic lymphocytic leukemia; stage II chronic lymphocytic leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; recurrent adult acute lymphoblastic leukemia; refractory chronic lymphocytic leukemia; untreated adult acute lymphoblastic leukemia; untreated childhood acute lymphoblastic leukemia; adult acute lymphoblastic leukemia in remission; childhood acute lymphoblastic leukemia in remission; untreated hairy cell leukemia; progressive hairy cell leukemia, initial treatment; refractory hairy cell leukemia; stage II childhood Hodgkin lymphoma; stage I childhood Hodgkin lymphoma; stage III childhood Hodgkin lymphoma; stage IV childhood Hodgkin lymphoma; recurrent/refractory childhood Hodgkin lymphoma; stage IV small lymphocytic lymphoma; stage I adult T-cell leukemia/lymphoma; stage II adult T-cell leukemia/lymphoma; stage III adult T-cell leukemia/lymphoma; stage IV adult T-cell leukemia/lymphoma; recurrent adult T-cell leukemia/lymphoma; stage I mycosis fungoides/Sezary syndrome; stage II mycosis fungoides/Sezary syndrome; stage III mycosis fungoides/Sezary syndrome; stage IV mycosis fungoides/Sezary syndrome; recurrent mycosis fungoides/Sezary syndrome; noncontiguous stage II small lymphocytic lymphoma; noncontiguous stage II marginal zone lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage I marginal zone lymphoma; stage I small lymphocytic lymphoma; stage II small lymphocytic lymphoma; stage II marginal zone lymphoma; stage III small lymphocytic lymphoma; stage III marginal zone lymphoma; stage IV marginal zone lymphoma; contiguous stage II marginal zone lymphoma; contiguous stage II small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Hodgkin Disease; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, T-Cell, Cutaneous; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Hairy Cell; Recurrence; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Mycosis Fungoides; Sezary Syndrome; Lymphoma, B-Cell, Marginal Zone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: allogeneic Epstein-Barr virus-specific cytotoxic T lymphocytes
Biological: autologous Epstein-Barr virus-specific cytotoxic T lymphocytes

SUMMARY:
RATIONALE: Peripheral blood lymphocyte therapy may be effective in the treatment and prevention of Epstein-Barr virus infection following transplantation.

PURPOSE: Phase II trial to study the effectiveness of peripheral blood lymphocyte therapy in treating and preventing lymphoproliferative disorders in patients who have Epstein-Barr virus infection following transplantation.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the efficacy of Epstein Barr virus (EBV) reactive autologous and allogeneic lymphocyte clones ex vivo in targeting EBV immortalized lymphoblasts in patients undergoing a solid organ transplant or T cell depleted bone marrow transplant.
* Determine the efficacy of these regimens as treatment and prophylaxis in those patients who develop EBV viremia or EBV induced lymphoproliferative disease.

OUTLINE: Autologous and allogeneic Epstein Barr virus (EBV) reactive lymphocytes are isolated from patients and siblings and tested in vitro for cytotoxic activity.

Patients who develop EBV viremia or EBV related lymphoproliferative disease after transplant receive autologous Epstein Barr virus (EBV) reactive lymphocytes IV over 20 minutes. Patients receive allogeneic EBV reactive lymphocytes if autologous lymphocytes fail to control EBV proliferation or when sufficient autologous reactive lymphocytes cannot be isolated. Treatment repeats every 4 weeks in the presence of EBV viremia or lymphoproliferative disease. After 5 patients have received therapy without unacceptable toxicity, patients may receive lymphocytes as prophylactic therapy.

Patients are followed at 4 weeks, 8 weeks, 6 months, and 12 months.

PROJECTED ACCRUAL: A total of 10-20 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Patients who have received or will receive a solid organ transplant or T cell depleted bone marrow transplant

  * Epstein Barr virus (EBV) DNA detectable and seronegative OR
  * EBV seropositive
* Fully matched or one HLA antigen mismatched sibling donor

  * HIV negative
  * Hepatitis B surface antigen negative
  * Hepatitis C antibody negative
  * No older than 65 years
  * No prior primary malignancy within the past 5 years in donor except previously resected skin cancer

PATIENT CHARACTERISTICS:

Age:

* Not specified

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2000-02; Primary Completion 2003-09 (Actual); Study Completion 2003-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ann Traynor, MD, Study Chair — Robert H. Lurie Cancer Center
Locations (1):
- Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois, United States